CLINICAL TRIAL: NCT02736266
Title: An Open Label, Single-arm, Phase 2 Study of Neoadjuvant Pembrolizumab (MK-3475) Before Cystectomy for Patients With Muscle-invasive Urothelial Bladder Cancer.
Brief Title: Neoadjuvant Pembrolizumab for Muscle-invasive Urothelial Bladder Carcinoma
Acronym: PURE-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Filippo de Braud, Prof., Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 101/16; 2015-002055-10 (EudraCT Number)
Record Dates: First submitted 2016-04-09; First posted 2016-04-13 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2022-11

CONDITIONS: Urothelial Bladder Carcinoma
Keywords: Muscle-invasive; Urothelial bladder carcinoma; Neoadjuvant therapy; Radical cystectomy
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (MK-3475) (Experimental): Pembrolizumab (MK-3475) will be administered at the dose of 200mg, as a 30-minute intravenous infusion, every 3 weeks, for a total of 3 cycles prior to radical cystectomy.
  Interventions: Drug: Pembrolizumab (MK-3475)

INTERVENTIONS:
Drug: Pembrolizumab (MK-3475) — Pembrolizumab given intravenously in 30 min. infusion every 3 weeks
  Other Names: Keytruda

SUMMARY:
Patients with T2-T4a N0 urothelial bladder carcinoma (UBC) with residual disease after transurethral resection of the bladder (TURB, surgical opinion, cystoscopy or radiological presence) will receive 3 cycles of pembrolizumab (MK-3475) at the dose of 200mg 3 weekly prior to surgery (radical cystectomy). Cystectomy will be planned to be done within 3 weeks of the last dose (accounting for a total of 9 weeks).

Computed tomography (CT) scan and fluorodeoxyglucose positron emission tomography (FDG-PET)/CT scan will be done during screening and before surgery. After cystectomy, patients with the evidence of pathologic stage T3-4 (pT3-4) and/or pathologically node-positive disease will be managed according to local guidelines. Further anti programmed-death (PD)-1 or anti PD-ligand 1 (PD-L1) therapy will not be given post-operatively.

PD-L1 status will be centralized and assessed on TURB specimen using an anti-PD-L1 antibody (Ab) and a prototype immunohistochemical (IHC) assay. PD-L1 positivity will be defined as any staining in the stroma or in ≥1% of tumor cells.

Pathologic complete response (pCR) is the primary endpoint. All patients enrolled who receive at least 1 cycle of study drug will be includes in the intention-to-treat (ITT) analysis.

The alternative hypothesis (H1) is pCR ≥20% and null hypothesis (H0) pCR≤10%. A 2-stage design will be used to estimate the number of pts required. Out of 90 pts overall, with the first stage of 49 pts, ≥6 pCR will be required in the first stage, and ≥13 pCR in the whole study population (80% power and a 2-sided test of significance at the 10% level).

Correlative research on tissue/blood samples will include immune-cell profiling in tumor and blood during Pembrolizumab, cytokine assessment, and molecular profiling of tumor samples.

DETAILED DESCRIPTION:
Patients with T2-T4a N0 urothelial bladder carcinoma (UBC) with residual disease after transurethral resection of the bladder (TURB, surgical opinion, cystoscopy or radiological presence) will receive 3 cycles of pembrolizumab (MK-3475) at the dose of 200mg 3 weekly prior to surgery (radical cystectomy). Cystectomy will be planned to be done within 3 weeks of the last dose (accounting for a total of 9 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Age ≥ 18 years.
4. Histopathologically confirmed transitional cell carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) transitional cell pattern.
5. Fit and planned for cystectomy (according to local guidelines).
6. Clinical stage T2-T4a N0 M0 disease by CT (or MRI) + PET/CT (within 4 weeks of randomization by RECIST v1.1).
7. Residual disease after TURB (surgical opinion, cystoscopy or radiological presence).
8. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens (blocks preferred) or at least 15 unstained slides, with an associated pathology report, for testing at the study sponsor site and determined to be evaluable for tumor PD-L1 expression prior to study enrolment; patients with fewer than 15 unstained slides available at baseline (but no fewer than 10) may be eligible following discussion with Merck representatives.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
10. Adequate hematologic and end-organ function tests.

Exclusion Criteria:

* Patients taking regular oral steroids, above the allowed limit of 10mg/day methylprednisolone or analogues, for any reason. Patients must not have had steroids for 28 days prior to study entry.
* Previously intravenous chemotherapy bladder cancer. Patients who have previously had radiotherapy or concurrent chemo-radiation would be eligible.
* Malignancies other than UBC within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
* Evidence of measurable nodal or metastatic disease.
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
* Pregnant female patients. All female patients of childbearing potential with a positive pregnancy test within 2 weeks prior to the first dose of study treatment will be excluded from the study.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias, or unstable angina.
* Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
* Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the pembrolizumab formulation
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Patients with a history of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
* Patients with uncontrolled Type 1 diabetes mellitus
* Uncontrolled hypercalcemia
* Patients with prior allogeneic stem cell or solid organ transplantation.
* History of idiopathic pulmonary fibrosis
* Positive test for HIV.
* Patients with active hepatitis infection
* Patients with active tuberculosis.
* Prior treatment with anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
* Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrolment
* History of severe immune-related adverse effects from anti-CTLA-4 (CTCAE Grade 3 and 4).
* Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response | At the time of radical cystectomy (within 9 weeks of the first dose of pembrolizumab)
  Absence of residual viable tumor in the radical cystectomy specimen

SECONDARY OUTCOMES:
Adverse events | Up to 2 years
  Number of patients developing side effects
Percentage of treatment-related delay in surgery | Starting at week 9
  Number of patients undergoing cystectomy later than 12 weeks after pembrolizumab treatment
Frequency of treatment-related adverse events | Up to 1 year
  Number of patients developing side effects

CONTACTS AND LOCATIONS:
Overall Officials: Filippo G. de Braud, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No
No formal plan

REFERENCES:
- [Derived] Necchi A, Basile G, Gibb EA, Raggi D, Calareso G, de Padua TC, Patane D, Crupi E, Mercinelli C, Cigliola A, Tateo V, Giannatempo P, Moschini M, Briganti A, Montorsi F, Messina A, Ross JS, Pavlick D, De Cobelli F, Brembilla G. Vesical Imaging-Reporting and Data System use predicting the outcome of neoadjuvant pembrolizumab in muscle-invasive bladder cancer. BJU Int. 2024 Feb;133(2):214-222. doi: 10.1111/bju.16191. Epub 2023 Oct 16. PMID 37803523
- [Derived] Basile G, Bandini M, Gibb EA, Ross JS, Raggi D, Marandino L, Costa de Padua T, Crupi E, Colombo R, Colecchia M, Luciano R, Nocera L, Moschini M, Briganti A, Montorsi F, Necchi A. Neoadjuvant Pembrolizumab and Radical Cystectomy in Patients with Muscle-Invasive Urothelial Bladder Cancer: 3-Year Median Follow-Up Update of PURE-01 Trial. Clin Cancer Res. 2022 Dec 1;28(23):5107-5114. doi: 10.1158/1078-0432.CCR-22-2158. PMID 36190522
- [Derived] Martini A, Raggi D, Marandino L, Montorsi F, Ross JS, Gibb EA, Necchi A. The Paradoxical Role of Body Mass Index in Patients with Muscle-invasive Bladder Cancer Receiving Neoadjuvant Immunotherapy. Eur Urol Oncol. 2022 Jun;5(3):370-372. doi: 10.1016/j.euo.2022.02.004. Epub 2022 Mar 10. No abstract available. PMID 35283158
- [Derived] Necchi A, Martini A, Raggi D, Cucchiara V, Colecchia M, Luciano R, Villa L, Mazzone E, Basile G, Scuderi S, Pederzoli F, Bandini M, Barletta F, Larcher A, Capitanio U, Salonia A, Briganti A, Ross JS, Messina A, Montorsi F. A feasibility study of preoperative pembrolizumab before radical nephroureterectomy in patients with high-risk, upper tract urothelial carcinoma: PURE-02. Urol Oncol. 2022 Jan;40(1):10.e1-10.e6. doi: 10.1016/j.urolonc.2021.05.014. Epub 2021 Jun 17. PMID 34147313
- [Derived] Trevisani F, Di Marco F, Raggi D, Bettiga A, Vago R, Larcher A, Cinque A, Salonia A, Briganti A, Capitanio U, Necchi A, Montorsi F. Renal function outcomes in patients with muscle-invasive bladder cancer treated with neoadjuvant pembrolizumab and radical cystectomy in the PURE-01 study. Int J Cancer. 2021 Jul 1;149(1):186-190. doi: 10.1002/ijc.33554. Epub 2021 Mar 26. PMID 33720424
- [Derived] Marandino L, Capozza A, Bandini M, Raggi D, Fare E, Pederzoli F, Gallina A, Capitanio U, Bianchi M, Gandaglia G, Fossati N, Colecchia M, Giannatempo P, Serafini G, Padovano B, Salonia A, Briganti A, Montorsi F, Alessi A, Necchi A. Incidence and Clinical Impact of Inflammatory Fluorodeoxyglucose Positron Emission Tomography Uptake After Neoadjuvant Pembrolizumab in Patients with Organ-confined Bladder Cancer Undergoing Radical Cystectomy. Eur Urol Focus. 2021 Sep;7(5):1092-1099. doi: 10.1016/j.euf.2020.10.003. Epub 2020 Nov 7. PMID 33172772
- [Derived] Marandino L, Capozza A, Bandini M, Raggi D, Fare E, Pederzoli F, Gallina A, Capitanio U, Bianchi M, Gandaglia G, Fossati N, Colecchia M, Giannatempo P, Serafini G, Padovano B, Salonia A, Briganti A, Montorsi F, Alessi A, Necchi A. [18F]Fluoro-Deoxy-Glucose positron emission tomography to evaluate lymph node involvement in patients with muscle-invasive bladder cancer receiving neoadjuvant pembrolizumab. Urol Oncol. 2021 Apr;39(4):235.e15-235.e21. doi: 10.1016/j.urolonc.2020.09.035. Epub 2020 Oct 16. PMID 33071107
- [Derived] Bandini M, Gibb EA, Gallina A, Raggi D, Marandino L, Bianchi M, Ross JS, Colecchia M, Gandaglia G, Fossati N, Pederzoli F, Luciano R, Colombo R, Salonia A, Briganti A, Montorsi F, Necchi A. Does the administration of preoperative pembrolizumab lead to sustained remission post-cystectomy? First survival outcomes from the PURE-01 study☆. Ann Oncol. 2020 Dec;31(12):1755-1763. doi: 10.1016/j.annonc.2020.09.011. Epub 2020 Sep 23. PMID 32979511
- [Derived] Pederzoli F, Bandini M, Marandino L, Raggi D, Giannatempo P, Salonia A, Gallina A, Briganti A, Montorsi F, Necchi A. Neoadjuvant Chemotherapy or Immunotherapy for Clinical T2N0 Muscle-invasive Bladder Cancer: Time to Change the Paradigm? Eur Urol Oncol. 2021 Dec;4(6):1006-1010. doi: 10.1016/j.euo.2020.07.006. Epub 2020 Aug 23. PMID 32847746
- [Derived] Bandini M, Calareso G, Raggi D, Marandino L, Colecchia M, Gallina A, Giannatempo P, Pederzoli F, Gandaglia G, Fossati N, Capitanio U, Colombo R, Salonia A, Briganti A, Montorsi F, De Cobelli F, Messina A, Necchi A. The Value of Multiparametric Magnetic Resonance Imaging Sequences to Assist in the Decision Making of Muscle-invasive Bladder Cancer. Eur Urol Oncol. 2021 Oct;4(5):829-833. doi: 10.1016/j.euo.2020.06.004. Epub 2020 Jun 27. PMID 32605888
- [Derived] Bandini M, Ross JS, Raggi D, Gallina A, Colecchia M, Luciano R, Giannatempo P, Fare E, Pederzoli F, Bianchi M, Colombo R, Gandaglia G, Fossati N, Marandino L, Capitanio U, Deho' F, Ali SM, Madison R, Chung JH, Salonia A, Briganti A, Montorsi F, Necchi A. Predicting the Pathologic Complete Response After Neoadjuvant Pembrolizumab in Muscle-Invasive Bladder Cancer. J Natl Cancer Inst. 2021 Jan 4;113(1):48-53. doi: 10.1093/jnci/djaa076. PMID 32516377
- [Derived] Necchi A, Raggi D, Giannatempo P, Marandino L, Fare E, Gallina A, Colecchia M, Luciano R, Salonia A, Gandaglia G, Fossati N, Bandini M, Pederzoli F, Dittamore R, Liu Y, Davicioni E, Ross JS, de Jong JJ, Briganti A, Montorsi F, Gibb EA. Can Patients with Muscle-invasive Bladder Cancer and Fibroblast Growth Factor Receptor-3 Alterations Still Be Considered for Neoadjuvant Pembrolizumab? A Comprehensive Assessment from the Updated Results of the PURE-01 Study. Eur Urol Oncol. 2021 Dec;4(6):1001-1005. doi: 10.1016/j.euo.2020.04.005. Epub 2020 May 14. PMID 32417369
- [Derived] Necchi A, Raggi D, Gallina A, Ross JS, Fare E, Giannatempo P, Marandino L, Colecchia M, Luciano R, Bianchi M, Colombo R, Salonia A, Gandaglia G, Fossati N, Bandini M, Pederzoli F, Capitanio U, Montorsi F, de Jong JJ, Dittamore R, Liu Y, Davicioni E, Boormans JL, Briganti A, Black PC, Gibb EA. Impact of Molecular Subtyping and Immune Infiltration on Pathological Response and Outcome Following Neoadjuvant Pembrolizumab in Muscle-invasive Bladder Cancer. Eur Urol. 2020 Jun;77(6):701-710. doi: 10.1016/j.eururo.2020.02.028. Epub 2020 Mar 9. PMID 32165065
- [Derived] Necchi A, Bandini M, Calareso G, Raggi D, Pederzoli F, Fare E, Colecchia M, Marandino L, Bianchi M, Gallina A, Colombo R, Fossati N, Gandaglia G, Capitanio U, Deho F, Giannatempo P, Luciano R, Salonia A, Madison R, Ali SM, Chung JH, Ross JS, Briganti A, Montorsi F, De Cobelli F, Messina A. Multiparametric Magnetic Resonance Imaging as a Noninvasive Assessment of Tumor Response to Neoadjuvant Pembrolizumab in Muscle-invasive Bladder Cancer: Preliminary Findings from the PURE-01 Study. Eur Urol. 2020 May;77(5):636-643. doi: 10.1016/j.eururo.2019.12.016. Epub 2019 Dec 25. PMID 31882281
- [Derived] Necchi A, Raggi D, Gallina A, Madison R, Colecchia M, Luciano R, Montironi R, Giannatempo P, Fare E, Pederzoli F, Bandini M, Bianchi M, Colombo R, Gandaglia G, Fossati N, Marandino L, Capitanio U, Deho F, Ali SM, Chung JH, Ross JS, Salonia A, Briganti A, Montorsi F. Updated Results of PURE-01 with Preliminary Activity of Neoadjuvant Pembrolizumab in Patients with Muscle-invasive Bladder Carcinoma with Variant Histologies. Eur Urol. 2020 Apr;77(4):439-446. doi: 10.1016/j.eururo.2019.10.026. Epub 2019 Nov 8. PMID 31708296
- [Derived] Necchi A, Montorsi F. Reply to S. Zhang. J Clin Oncol. 2019 Apr 10;37(11):940-941. doi: 10.1200/JCO.18.02448. Epub 2019 Feb 27. No abstract available. PMID 30811283
- [Derived] Necchi A, Anichini A, Raggi D, Briganti A, Massa S, Luciano R, Colecchia M, Giannatempo P, Mortarini R, Bianchi M, Fare E, Monopoli F, Colombo R, Gallina A, Salonia A, Messina A, Ali SM, Madison R, Ross JS, Chung JH, Salvioni R, Mariani L, Montorsi F. Pembrolizumab as Neoadjuvant Therapy Before Radical Cystectomy in Patients With Muscle-Invasive Urothelial Bladder Carcinoma (PURE-01): An Open-Label, Single-Arm, Phase II Study. J Clin Oncol. 2018 Dec 1;36(34):3353-3360. doi: 10.1200/JCO.18.01148. Epub 2018 Oct 20. PMID 30343614